CLINICAL TRIAL: NCT05556382
Title: Glioblastoma Evaluation for Heterogeneity In RadioseNsitivity (GEHIRN): Preclinical Observational Study on Ex-vivo Surgical Specimens
Brief Title: Glioblastoma Evaluation for Heterogeneity In RadioseNsitivity
Acronym: GEHIRN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 3075
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh brain tissue sample witdraw during tumor surgical resection. Tissue samples will be incubated in culture medium for 24 hours and exposed to increasing single radiation dose (0, 2, 4, 6 Gy) with a linear accelerator. Specimens will be further incubated for 24 hours and subsequently fixed in formaldehyde and paraffin-embedded: γH2AX analysis will be conducted on cross-sections from the paraffin-embedded tumor material after tissue staining using confocal microscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: radiation of brain tissue specimen and dna damage analysis — increasing doses of radiation on brain tissue specimen and analysis of related dna damage.

SUMMARY:
This is an observational study on GBM surgical samples to investigate if increasing doses of radiation therapy could improve the radiation response; and in particular the investigators will assess if there is a correlation between the number of the phosphorylated H2AX nuclear foci and the different dose level of radiation therapy.

DETAILED DESCRIPTION:
Standard of care for newly diagnosed glioblastoma (GBM) patients consists of surgical resection followed by radiotherapy with concurrent and adjuvant Temozolomide chemotherapy. Despite these treatments, the prognosis remains poor. Nevertheless, preliminary data on GBM patients show variable outcomes related to a different treatment response, that could be related to the GBM intrinsic heterogeneity, but also to a different patient sensitivity to radiation therapy.

The assessment of this individual radio-sensitivity may provide valuable data to define more tailored treatment schedules, that could potentially be more effective.

Published studies on small cohort of patients show that a possible system to investigate the tumor radiation sensitivity, is to monitor the cellular DNA damage after tissue irradiation, that correlates with the survival fraction of in vitro tumor cells; the DNA damage could be identified through the quantification of Phosphorylated histone H2AX nuclear foci that correlate with the unrepaired DNA double strand breaks (DSBs).

Based on this background, The investigators designed an observational study on GBM surgical samples to investigate if increasing doses of radiation therapy could improve the radiation response; and in particular they will assess if there is a correlation between the number of the phosphorylated H2AX nuclear foci and the different dose level of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years
* Patients eligible for diagnostic or therapeutic surgical procedure
* Written informed consent
* Histopathologically confirmed newly diagnosed glioblastoma according to WHO 2021
* Availability of fresh tissue samples

Exclusion Criteria:

* Other extra-cranial cancer
* Non GBM glioma
* Previous brain radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioblastoma Patients eligible for surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Determination of distribution of number of γH2AX foci in each irradiated specimen (Nfoci) for each radiation dose level | 1 month
  Number of foci per irradiated sample (Nfoci) for each dose level expressed as [(number of observed γH2AX foci per selected dose level)-(number of observed γH2AX foci in control unirradiated sample)].

SECONDARY OUTCOMES:
correlation between n° of γH2AX foci and dose levels | 1 month
  this correlation will be described by the slope for each sample Nfoci at increasing dose levels

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Clinical Institute, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided